CLINICAL TRIAL: NCT04662567
Title: Oral Versus Intravenous Acetaminophen for Postoperative Pain Management After Oocyte Retrieval Procedure. A Double Blinded, Placebo Controlled, Randomized Clinical Trial
Brief Title: Oral Versus Intravenous Acetaminophen for Postoperative Pain Control
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: It was determined that the study should not continue as the study drug, Acetaminophen, could only be mixed in a solvent that would not allow the patients to be NPO prior to procedure.
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 20-1139
Record Dates: First submitted 2020-11-16; First posted 2020-12-10 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Postoperative Pain; IVF
Keywords: oocyte retrieval; postoperative pain control; in vitro fertilization; tylenol
MeSH Terms: conditions — Pain, Postoperative | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oral acetaminophen group (Active Comparator): the subjects in this group will receive 1000 mg oral acetaminophen 30-45min prior to oocyte retrieval
  Interventions: Drug: acetaminophen
- IV acetaminophen group (Active Comparator): the subjects in this group will receive 1000 mg IV acetaminophen formulation intraoperatively
  Interventions: Drug: acetaminophen

INTERVENTIONS:
Drug: acetaminophen — compare the postoperative pain 1 hour and ~24h post surgery

SUMMARY:
The investigators are going to study the difference in postoperative pain control after administration of oral versus intravenous formulation of acetaminophen

DETAILED DESCRIPTION:
Oocyte retrieval is an outpatient procedure that is a routine surgical intervention in the process of assisted reproductive technologies and oocyte banking. The perioperative pain control is achieved with multidrug regimen including intraoperative opioid medication and perioperative administration of oral or intravenous acetaminophen. This medication is more commonly known as Tylenol. Intravenous formulation of this medication is several fold more expensive and the data for perioperative pain control is mixed on the equivalence of pain control with intravenous versus oral acetaminophen in other fields. Currently there is no accepted standard of care and the two formulations are used interchangeably depending on primary physician's preference. We are conducting an equivalence placebo controlled randomized clinical trial to assess the difference in efficacy of these two formulations

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Female, aged 18-45
4. Ability to take oral medication and be willing to adhere to the study intervention regimen

Exclusion Criteria:

1. Known clinically significant liver disfunction
2. Known allergic reactions to components of acetaminophen such as angioedema, anaphylaxis or other
3. Known current substance use disorder
4. Chronic pain syndrome
5. Weight less than 50 kg

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2021-03-12 (Actual); Primary Completion 2021-09-05 (Actual); Study Completion 2021-09-05 (Actual)

PRIMARY OUTCOMES:
postoperative pain control | 24-48 hours
  To compare the efficacy of oral versus IV formulation of acetaminophen for controlling perioperative pain after oocyte retrieval procedure.
  To assess the pain level, Visual Analog Scale(VAS) score will be utilize with the minimum number 0 representing no pain and maximum number of 10 representing the highest imaginable pain level.

SECONDARY OUTCOMES:
Duration of postoperative recovery | variable ~1-3 hours
  To compare time from the end of procedure until discharge. This outcome is measured in minutes from the the time of entry to recovery room to the time when patient is leaving the facility

CONTACTS AND LOCATIONS:
Overall Officials: Christine Mullin, MD, Principal Investigator — Northwell Health OBGYN Infertility
Locations (1):
- Northwell Fertility Center #3816, Manhasset, New York, United States

IPD SHARING:
Plan to Share IPD: No
the individual participant data will not be shared

REFERENCES:
- [Background] Alloui A, Chassaing C, Schmidt J, Ardid D, Dubray C, Cloarec A, Eschalier A. Paracetamol exerts a spinal, tropisetron-reversible, antinociceptive effect in an inflammatory pain model in rats. Eur J Pharmacol. 2002 May 17;443(1-3):71-7. doi: 10.1016/s0014-2999(02)01578-9. PMID 12044794
- [Background] Flower RJ, Vane JR. Inhibition of prostaglandin synthetase in brain explains the anti-pyretic activity of paracetamol (4-acetamidophenol). Nature. 1972 Dec 15;240(5381):410-1. doi: 10.1038/240410a0. No abstract available. PMID 4564318
- [Background] Graham GG, Scott KF. Mechanism of action of paracetamol. Am J Ther. 2005 Jan-Feb;12(1):46-55. doi: 10.1097/00045391-200501000-00008. PMID 15662292
- [Background] Hinz B, Brune K. Paracetamol and cyclooxygenase inhibition: is there a cause for concern? Ann Rheum Dis. 2012 Jan;71(1):20-5. doi: 10.1136/ard.2011.200087. Epub 2011 Oct 28. PMID 22039164
- [Background] Hinz B, Cheremina O, Brune K. Acetaminophen (paracetamol) is a selective cyclooxygenase-2 inhibitor in man. FASEB J. 2008 Feb;22(2):383-90. doi: 10.1096/fj.07-8506com. Epub 2007 Sep 20. PMID 17884974
- [Background] Hinz B, Dormann H, Brune K. More pronounced inhibition of cyclooxygenase 2, increase in blood pressure, and reduction of heart rate by treatment with diclofenac compared with celecoxib and rofecoxib. Arthritis Rheum. 2006 Jan;54(1):282-91. doi: 10.1002/art.21540. PMID 16385545
- [Background] Jahr JS, Lee VK. Intravenous acetaminophen. Anesthesiol Clin. 2010 Dec;28(4):619-45. doi: 10.1016/j.anclin.2010.08.006. PMID 21074742
- [Background] Moller PL, Sindet-Pedersen S, Petersen CT, Juhl GI, Dillenschneider A, Skoglund LA. Onset of acetaminophen analgesia: comparison of oral and intravenous routes after third molar surgery. Br J Anaesth. 2005 May;94(5):642-8. doi: 10.1093/bja/aei109. Epub 2005 Mar 24. PMID 15790675
- [Background] Nakamura K, Li YQ, Kaneko T, Katoh H, Negishi M. Prostaglandin EP3 receptor protein in serotonin and catecholamine cell groups: a double immunofluorescence study in the rat brain. Neuroscience. 2001;103(3):763-75. doi: 10.1016/s0306-4522(01)00027-6. PMID 11274793
- [Background] Pasero C, Stannard D. The role of intravenous acetaminophen in acute pain management: a case-illustrated review. Pain Manag Nurs. 2012 Jun;13(2):107-24. doi: 10.1016/j.pmn.2012.03.002. PMID 22652283
- [Background] Pickering G, Esteve V, Loriot MA, Eschalier A, Dubray C. Acetaminophen reinforces descending inhibitory pain pathways. Clin Pharmacol Ther. 2008 Jul;84(1):47-51. doi: 10.1038/sj.clpt.6100403. Epub 2007 Oct 24. PMID 17957182
- [Background] Pickering G, Loriot MA, Libert F, Eschalier A, Beaune P, Dubray C. Analgesic effect of acetaminophen in humans: first evidence of a central serotonergic mechanism. Clin Pharmacol Ther. 2006 Apr;79(4):371-8. doi: 10.1016/j.clpt.2005.12.307. PMID 16580905